CLINICAL TRIAL: NCT04635592
Title: Serological Diagnostics of COVID-19 and Risk Factors for Infection Among Different Groups of Health Care Workers at Surgical Division at Tertiary Hospital
Brief Title: Serological Diagnostics of COVID-19 in Health Care Workers
Acronym: KORANIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Peter Poredos, Assist. prof., University Medical Centre Ljubljana
Other Study IDs: KOAIT-1-2020
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: SARS-CoV Infection
Keywords: SARS-CoV2 infection; Health care worker; Serology; Nasal swab tests; Anesthesiology and Intensive Care
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SARS-CoV2 nasal swabs Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV2 nasal swab — SARS-CoV2 nasal swab and venous blood for SARS-CoV2 antibodies

SUMMARY:
All health care workers at the Department of Anesthesiology and Intensive Care at UMC Ljubljana will be tested for SARS-CoV2 with nasal swab test and blood withdrawal for SARS-CoV2 antibodies. At the same time a questionnaire with epidemiological anamnesis, risky contacts and the use of personal protective equipment will be fulfilled.

DETAILED DESCRIPTION:
Health care workers at the Department of Anesthesiology and Intensive Care at UMC Ljubljana are working with COVID-19 patients in intensive care units, operating theaters, wards and emergency department. In the care of those patients different workgroups are involved: anesthesiologists, anesthesia and ICU nurses and respiratory therapeuts.There is insufficient data on the seroprevalence in different workgroups, different areas of the hospital, insufficient data on connection between SARS-CoV2 nasal swabs and antibodies and the rate of asymptomatic infections.

300 hundred HCW will be tested for SARS-CoV2 with nasal swab test and blood withdrawal for SARS-CoV2 antibodies. At the same time a questionnaire with epidemiological anamnesis, risky contacts and the use of personal protective equipment will be filled.

ELIGIBILITY:
Inclusion Criteria:

* employee of Department of Anesthesiology and Intensive Care at UMC Ljubljana
* active current employment at the department

Exclusion Criteria:

* current sick-leave

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers at Department of Anesthesiology and Intensive Care at UMC Ljubljana
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
positive nasal swab and serological test | 2 months
  Rate of positive nasal swab and serological tests for SARS-CoV2 among health care workers

SECONDARY OUTCOMES:
Relation of positive SARS-CoV2 tests to risky contact history | 8 months
  Relation of positive SARS-CoV2 tests to history of contacts with COVID-19 infected patients since the beginning of pandemia

CONTACTS AND LOCATIONS:
Overall Officials: Peter Poredos, MD, PhD, Study Chair — Department of Anesthesiology and Intensive Care - Hear
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Basteiro AL, Moncunill G, Tortajada M, Vidal M, Guinovart C, Jimenez A, Santano R, Sanz S, Mendez S, Llupia A, Aguilar R, Alonso S, Barrios D, Carolis C, Cistero P, Choliz E, Cruz A, Fochs S, Jairoce C, Hecht J, Lamoglia M, Martinez MJ, Mitchell RA, Ortega N, Pey N, Puyol L, Ribes M, Rosell N, Sotomayor P, Torres S, Williams S, Barroso S, Vilella A, Munoz J, Trilla A, Varela P, Mayor A, Dobano C. Seroprevalence of antibodies against SARS-CoV-2 among health care workers in a large Spanish reference hospital. Nat Commun. 2020 Jul 8;11(1):3500. doi: 10.1038/s41467-020-17318-x. PMID 32641730
- [Background] Rudberg AS, Havervall S, Manberg A, Jernbom Falk A, Aguilera K, Ng H, Gabrielsson L, Salomonsson AC, Hanke L, Murrell B, McInerney G, Olofsson J, Andersson E, Hellstrom C, Bayati S, Bergstrom S, Pin E, Sjoberg R, Tegel H, Hedhammar M, Phillipson M, Nilsson P, Hober S, Thalin C. SARS-CoV-2 exposure, symptoms and seroprevalence in healthcare workers in Sweden. Nat Commun. 2020 Oct 8;11(1):5064. doi: 10.1038/s41467-020-18848-0. PMID 33033249
- [Background] Oran DP, Topol EJ. Prevalence of Asymptomatic SARS-CoV-2 Infection : A Narrative Review. Ann Intern Med. 2020 Sep 1;173(5):362-367. doi: 10.7326/M20-3012. Epub 2020 Jun 3. PMID 32491919
- [Background] Gomez-Ochoa SA, Franco OH, Rojas LZ, Raguindin PF, Roa-Diaz ZM, Wyssmann BM, Guevara SLR, Echeverria LE, Glisic M, Muka T. COVID-19 in Health-Care Workers: A Living Systematic Review and Meta-Analysis of Prevalence, Risk Factors, Clinical Characteristics, and Outcomes. Am J Epidemiol. 2021 Jan 4;190(1):161-175. doi: 10.1093/aje/kwaa191. PMID 32870978